CLINICAL TRIAL: NCT02514993
Title: The Unstable Thoracic Cage Injury: The Concomitant Sternal Fracture Indicates a Severe Thoracic Spine Fracture
Brief Title: The Unstable Thoracic Cage Injury
Status: Completed | Type: Observational
Sponsor: BG Unfallklinik Murnau (Other)
Responsible Party: Principal Investigator, Dr. Mario Morgenstern, M.D., BG Unfallklinik Murnau
Other Study IDs: 10-2004-2013
Record Dates: First submitted 2015-07-31; First posted 2015-08-04 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Thoracic Spine Fracture; Concomitant Sternal Fracture
Keywords: Sternal fracture; Thoracic spine fracture; Thoracic cage injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study group: Inclusion criteria for the study were (a) sternal fracture and concomitant thoracic spine fracture, (b) Injury Severity scale (ISS) ≥ 16, (c) age under 50 years, (d) presence of a whole body computed-tomography (CT-scan) performed at admission of the patient to the hospital.
- Control group: The inclusion criteria for the control group included: (a) Thoracic spine fracture without concomitant sternal fracture, (b) ISS ≥ 16, (c) age under 50 years, (d) presence of a whole body computed-tomography (CT-scan) performed at admission of the patient to the hospital.

SUMMARY:
* Analysis of patient data and computed tomography scan of polytraumatized patients thoracic spine fractures
* A concomitant sternal fracture was identified an indicator for an unstable thoracic spine fracture

DETAILED DESCRIPTION:
Previous studies stated, that sternal fractures can be regarded as an indicator for thoracic spine fractures and described the combined injury pattern of thoracic spine fracture and sternal fracture as "upper thoracic cage injury". But literature research is lacking data that in patients with a thoracic cage injury a highly unstable thoracic spine fracture can be expected.

In a large cohort of 130 patients with a thoracic spine fracture and concomitant sternal fracture the investigators analyzed the injury pattern and evaluated associated injuries, trauma mechanism, and clinical outcome.

The investigators could prove that in patients with a thoracic cage injury the concomitant sternal fracture may be regarded as an indicator for an unstable thoracic spine fracture, which requires surgical stabilization. Furthermore the analysis revealed that even a highly rotationally unstable type C fracture has to be expected, if sternal and thoracic spine fractures are located in the same segment.

ELIGIBILITY:
Inclusion Criteria:

* Sternal fracture and concomitant thoracic spine fracture
* Injury Severity Scale ≥ 16
* Age under 50 years
* Presence of a whole body computed-tomography (CT-scan) performed at admission of the patient to the hospital

Exclusion Criteria:

* Missing consent
* Incomplete patient data

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients suffering a thoracic spine fracture and a concomitant sternal fracture
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2003-01; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Survival | 1 year after trauma
  Patient survival after polytraumatization

CONTACTS AND LOCATIONS:
Overall Officials: Mario Morgenstern, M.D., Principal Investigator — Trauma Center Murnau